CLINICAL TRIAL: NCT05236296
Title: Pilot Study of a Novel Psychotherapeutic Intervention for Caregivers of Patients With Acute Leukemia: Emotion and Symptom-focused Engagement for Caregivers (EASE-CG)
Brief Title: Emotion and Symptom-focused Engagement for Caregivers (EASE-CG) Pilot Study
Acronym: EASE-CG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-5452
Record Dates: First submitted 2022-02-01; First posted 2022-02-11 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Leukemia, Acute
Keywords: Caregivers; Psychosocial Intervention; Traumatic Stress; Hematological Malignancies; Supportive Care; Acute Leukemia
MeSH Terms: conditions — Leukemia; Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: All study participants will receive the EASE-CG intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EASE-CG Intervention (Experimental): Participants will be offered one EASE-CG therapy session every week for up to 12 weeks. Each session will last for approximately 30-60 minutes, delivered by a trained therapist at our center. Frequency and/or length of sessions may vary to accommodate the needs and availability of each participant.
  Outcomes will be assessed at baseline, 1, 3, 6, 9, and 12 months. Participants may be invited to brief, semi-structured interviews.
  Interventions: Behavioral: EASE-CG

INTERVENTIONS:
Behavioral: EASE-CG — EASE-CG is an adapted brief psychotherapeutic intervention with relational support and trauma-based cognitive behavioral therapy (CBT) components.

SUMMARY:
The purpose of this study is to test the feasibility and acceptability of an adapted psychosocial intervention, called Emotion and Symptom-focused Engagement for Caregivers (EASE-CG), to reduce traumatic stress symptoms and other psychological distress and increase well-being in primary caregivers of patients newly diagnosed with acute leukemia.

DETAILED DESCRIPTION:
Emotion and Symptom-focused Engagement for Caregivers (EASE-CG) is a brief psychotherapeutic intervention designed for primary caregivers of patients newly diagnosed with acute leukemia (AL). The EASE-CG intervention was adapted from a previous psychotherapeutic intervention for adult patients newly diagnosed with AL, called Emotion and Symptom-focused Engagement (EASE). In a previous pilot trial, EASE was associated with reductions in traumatic stress and physical symptom burden in adult patients with AL.

EASE-CG is a sub-study of a multi-center, longitudinal, mixed-methods study on the experience of traumatic stress in primary caregivers of patients newly diagnosed with AL within three months of admission to the hospital (Main study). The purpose of this sub-study is to conduct a non-randomized, mixed-methods pilot study to test the feasibility and acceptability of EASE-CG. A subset of caregivers of pediatric patients from the Main study will be approached to participate in EASE-CG. Quantitative measures will be administered at baseline, 1, 3 (primary endpoint), 6, 9, and 12 months (Main study endpoint). Participants may be invited to brief, semi-structured interviews.

The study will take place at the Hospital for Sick Children; the largest leukemia treatment center in Canada for pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified primary caregiver (i.e., person assuming the majority of care activities) or co-primary caregiver (i.e., assuming at least 40% of care activities alongside another co-primary caregiver) of an adult or pediatric patient who is newly diagnosed with acute leukemia within 3 months of admission to the Princess Margaret Cancer Centre or the Hospital for Sick Children
* Age ≥18 years
* Fluency in English

Exclusion Criteria: none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Stanford Acute Stress Reaction Questionnaire (SASRQ-II) | 12 weeks
  A 30-item reliable, valid, and widely used self-report measure assessing the severity of traumatic stress symptoms over the past four weeks. Total SASRQ scores may range from 0-150, with higher scores indicating increasingly severe traumatic stress symptoms. This measure has been updated to be Diagnostic and Statistical Manual of Mental Disorders (DSM-5)-concordant for acute stress disorder symptoms.
PTSD Checklist for DSM-5 (PCL-5) | 12 weeks
  A 20-item reliable and valid self-report measure of the presence and severity of post-traumatic stress disorder (PTSD) symptoms over the past month. Total PCL-5 scores may range from 0-80, with higher scores indicating increasingly severe PTSD symptoms. This DSM-5-concordant measure has been included to help validate the DSM-5-concordant version of the SASRQ.

SECONDARY OUTCOMES:
Brief Experiences in Close Relationships Scale (ECR-M16) | 12 weeks
  A 16-item reliable and valid self-report measure of attachment security (i.e., the ability to rely on close others for support when distressed); in addition to a total score, it has subscales assessing anxious and avoidant attachment. Total ECR-M16 scores may range from 16-112, with higher scores indicating poorer attachment security (or greater attachment insecurity).
Patient Health Questionnaire-9 (PHQ-9) | 12 weeks
  A 9-item reliable and valid measure of depressive symptoms that has been widely used in patients with cancer. Total PHQ-9 scores may range from 0-27, with higher scores indicating increasingly severe depressive symptoms.
Caregiver Reaction Assessment (CRA) Scale | 12 weeks
  A 24-item reliable and valid measure of the positive and negative reactions to five dimensions of caregiver burden: (1) impact on schedule (i.e., disruption to usual daily activities) (5 items), (2) impact on finances (i.e., financial strain) (3 items), (3) lack of family support (5 items), (4) impact on caregiver's health (4 items), and (5) impact on caregiver's self-esteem (7 items). Higher scores indicate a stronger impact of caregiving on each dimension (either negative or positive). For dimensions 1-4, higher scores indicate higher negative experiences of caregiving. For dimension 5, higher scores indicate a higher level of positive caregiving experience. No overall summed score is used.
Enhancing Recovery In Coronary Heart Disease (ENRICHD) Social Support Inventory (ESSI) | 12 weeks
  A 7-item reliable and valid measure of the perceived availability of social support. Total ESSI scores may range from 6-31, with higher scores indicating greater perceived social support.
Family Satisfaction with End-of-Life Care (FAMCARE) Scale | 12 weeks
  A 20-item reliable and valid measure of satisfaction with health care practitioners' behaviour towards family caregivers and their loved ones with advanced cancer. Total FAMCARE scores may range from 20-100, with higher scores indicating greater caregiver satisfaction with health care practitioners.
Traditional Masculinity-Femininity (TMF) Scale | Baseline
  A 6-item reliable and valid measure of gender role, or the extent to which people view their interests, behaviour, attitudes and other aspects of themselves as masculine or feminine. Total TMF scores may range from 6-42, with higher scores indicating a greater sense of femininity. A score of four indicates an equal balance between masculine and feminine traits.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Rodin, MD FRCPC, Principal Investigator — University Health Network, Toronto; Lindsay Jibb, RN PhD, Principal Investigator — The Hospital for Sick Children
Locations (2):
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

REFERENCES:
- [Background] Rodin G, Malfitano C, Rydall A, Schimmer A, Marmar CM, Mah K, Lo C, Nissim R, Zimmermann C. Emotion And Symptom-focused Engagement (EASE): a randomized phase II trial of an integrated psychological and palliative care intervention for patients with acute leukemia. Support Care Cancer. 2020 Jan;28(1):163-176. doi: 10.1007/s00520-019-04723-2. Epub 2019 Apr 17. PMID 31001692
- [Derived] Jibb LA, Yu A, Nanos S, Malfitano C, Foran L, Hunt K, Malakian A, Zimmermann C, Schultebraucks K, Pham NA, Rydall A, Alexander S, Rodin G. The Emotion and Symptom-Focused Engagement (EASE) Psychotherapeutic Intervention for Parents of Children With Acute Leukemia: A Feasibility Trial. Psychooncology. 2025 Nov;34(11):e70310. doi: 10.1002/pon.70310. PMID 41161769